CLINICAL TRIAL: NCT01423461
Title: Individualized Health Care for Children With Common Chronic Diseases
Brief Title: Personalized Asthma Care Team
Acronym: PACT
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: The Cleveland Foundation (Other); University Hospitals Cleveland Medical Center (Other); Case Western Reserve University (Other); National Center for Research Resources (NCRR) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Susan Redline, Senior Physician, Division of Sleep Medicine, Brigham and Women's Hospital
Other Study IDs: L2005-0254; KL2RR024990 (NIH); UL1RR024989 (NIH); 1U54CA116867 (NIH); M01RR000080 (NIH)
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Asthma; Sleep Disordered Breathing; Obesity
MeSH Terms: conditions — Asthma; Sleep Apnea Syndromes; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
"Individualized health care" refers to the development of strategies for disease management and health promotion that are informed by specific data on genetics and physiological processes that uniquely determine each person's health profile and potential responsiveness to interventions or susceptibility to environmental exposures.

Asthma, an inflammatory disorder of the airway, appears to be determined by multiple interacting genetic and environmental factors. Such risk factors include allergic responses, small airways, excess body weight, specific properties of airway smooth muscle, airway and generalized metabolic and inflammatory homeostasis, and exposures to environmental irritants, allergens, and psychosocial stressors. To date, asthma treatment strategies have been guided by "severity" guidelines rather than by characteristics of the child's specific phenotype (a child's underlying allergic tendency, extent of airway inflammation and airway smooth muscle dysfunction, or underlying obesity and metabolic perturbations). The growing availability of new classes of asthma medications that more directly target specific pathophysiological derangements will require accessing data on each child's asthma risk profiles to optimize selection of medications and other interventions that most specifically address the underlying pathophysiology while minimizing adverse treatment side effects.

The investigators propose to develop a model program for collecting relevant clinical information and genetic data on a high risk group of asthmatic children, including data on common co-morbidities, specifically obesity and sleep disorders; use this information to develop a comprehensive model database for characterizing children according to their health profiles; and use this characterization to initiate targeted interventions, while continuing long term follow up of these children to determine differential responsiveness to medications.

ELIGIBILITY:
Inclusion Criteria:

* ages 4 to 18 years
* diagnosis of asthma or symptoms of persistent wheeze, unexplained by an etiology other than asthma

Exclusion Criteria:

* other severe co-morbidity (cystic fibrosis, sickle cell disease, chronic lung disease of prematurity, interstitial lung disease, cerebral palsy)
* inability of family to provide informed consent
* plans of the family to move out of the greater Cleveland area in the subsequent 24 months
* or inability to participate in regular follow up visits

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children seen at the pediatric pulmonology department with a diagnosis of asthma or symptoms of persistent wheeze, unexplained by an etiology other than asthma, ages 4 to 18 years will be recruited.
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2005-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Redline, M.D., M.P.H., Study Director — Brigham and Women's Hospital; Kristie Ross, M.D., Principal Investigator — University Hospitals Cleveland Medical Center; Meeghan Hart, M.D., Principal Investigator — University Hospitals Cleveland Medical Center; Carol Rosen, M.D., Principal Investigator — University Hospitals Cleveland Medical Center